CLINICAL TRIAL: NCT02007655
Title: Eliquis Safety Surveillance in Japanese Patients With NonValvular Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-286
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: NonValvular Atrial Fibrillation
Keywords: Cardiovascular
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Eliquis on Nonvalvular Atrial Fibrilliation patients: Patients who are beginning to receive the treatment with Eliquis under the approved indications, dosage, and administration will be included in this study
  Interventions: Drug: Eliquis

INTERVENTIONS:
Drug: Eliquis
  Other Names: Apixaban; BMS-562247

SUMMARY:
The primary objectives of this study are:

* To estimate the incidence rate of unexpected adverse events
* To characterize the bleeding events and assess risk factors of bleeding
* To identify ancillary baseline variables that may also be associated with adverse outcomes

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Patients who are beginning to receive the treatment with this product under the approved indications, dosage, and administration will be included in this study

Exclusion Criteria:

* Patients who are receiving Eliquis outside of its approved indication will be excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University hospitals, general hospitals, and clinics that have relevant departments, such as cardiology, cerebrovascular medicine, neurology, internal medicine, neurosurgery, etc, where the surveillance drug is mainly prescribed
Sampling Method: Non-Probability Sample
Enrollment: 6372 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of unexpected adverse events | Day 1 (At Eliquis initiation)
Incidence rate of unexpected adverse events | 12 weeks after initiation
Incidence rate of unexpected adverse events | 52 weeks after initiation
Incidence rate of unexpected adverse events | 104 week (discontinuation)
Bleeding events and risk factors of bleeding | Day 1 (At Eliquis initiation)
Bleeding events and risk factors of bleeding | 12 weeks after initiation
Bleeding events and risk factors of bleeding | 52 weeks after initiation
Bleeding events and risk factors of bleeding | 104 week (discontinuation)
Ancillary baseline variables that may also be associated with adverse outcomes | Day 1 (At Eliquis initiation)
Ancillary baseline variables that may also be associated with adverse outcomes | 12 weeks after initiation
Ancillary baseline variables that may also be associated with adverse outcomes | 52 weeks after initiation
Ancillary baseline variables that may also be associated with adverse outcomes | 104 week (discontinuation)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Toyama, Toyama, Japan

REFERENCES:
- [Derived] Inoue H, Umeyama M, Yamada T, Hashimoto H, Komoto A, Yasaka M. Safety and effectiveness of reduced-dose apixaban in Japanese patients with nonvalvular atrial fibrillation in clinical practice: A sub-analysis of the STANDARD study. J Cardiol. 2020 Feb;75(2):208-215. doi: 10.1016/j.jjcc.2019.07.007. Epub 2019 Aug 15. PMID 31421933
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm